CLINICAL TRIAL: NCT01454154
Title: A Randomized Clinical Trial of Glyburide (RP-1127) for TBI
Brief Title: Glyburide (RP-1127) for Traumatic Brain Injury (TBI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Remedy Pharmaceuticals, Inc. (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPI 202; INTRuST-GLY (Other: INTRuST Clinical Consortium Coordinating Center)
Record Dates: First submitted 2011-10-11; First posted 2011-10-18 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glyburide (Experimental): Glyburide delivered by injection as an approximately 2 minute loading dose followed by 72 hours of continuous infusion.
  Interventions: Drug: Glyburide
- Placebo (Placebo Comparator): Matching placebo delivered by injection as an approximately 2 minute loading dose followed by 72 hours of continuous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glyburide — Administered as specified in the Treatment Arm.
  Other Names: RP-1127; glibenclamide; glybenclamide
  Arms: Glyburide
Drug: Placebo — Administered as specified in the Treatment Arm.
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to assess whether participants with traumatic brain injury (TBI) administered glyburide begun within 10 hours of injury will show a decrease in magnetic resonance imaging (MRI)-defined edema and/or hemorrhage, compared to placebo and to assess the safety and tolerability of glyburide compared to placebo in participants with TBI. The secondary objectives include analyzing brain cell loss, computerized tomography (CT) scan /MRI abnormalities, reduction of mortality and or improvement of function or physiology, incidence of decompression craniectomy, incidence of neuroworsening, and to assess the steady state concentrations of glyburide in TBI participants.

ELIGIBILITY:
Inclusion Criteria:

1. Documented closed head TBI
2. Clearly defined time of injury no more than 10 hours before administration of study drug/placebo
3. GCS 4-14. The GCS will be obtained free of the effects of sedating and/or paralytic drug. Complicated mild must have GCS 13-14 and one or more of the following: Intraparenchymal clots or contusions in aggregate > 10cc; Midline shift > 5mm; IVH, SDH, EDH seen on more than one CT scan slice.
4. Age 18-75 years
5. Patients in whom a dedicated peripheral IV line can be placed for study drug administration
6. Written consent obtained from legally authorized representative (LAR)

Exclusion Criteria:

1. No documented TBI or time of impact not certain
2. Penetrating brain injury
3. Spinal column instability and/or spinal cord injury with neurodeficit
4. Concomitant severe non survivable injury
5. Pregnant, or a positive pregnancy test
6. Women who intend to breastfeed during Study Days 1-4.
7. Blood glucose <50mg/dL
8. Severe renal disorder from the patient's history (e.g. dialysis) or serum creatinine of > 2.5 mg/dL
9. Severe liver disease or total bilirubin >1.5 times upper limit of normal
10. INR>1.4
11. Systolic BP<90 mm Hg not responsive to fluid resuscitation
12. Blood alcohol > 250mg/dL
13. Inability to have MRI (pacemaker, non-MR compatible pressure monitor, etc.)
14. Hospitalization for brain injury, psychiatric or neurological disease within previous 3 years
15. Emergent or urgent surgical operation anticipated (in OR, bedside procedures excluded) that would prevent dosing with study drug within 8 hours of injury.
16. Known use of Coumadin (warfarin), Plavix (clopidogrel), Effient (prasugrel) or Pletal (cilostazol), heparin, low molecular weight heparin, heparinoids, or abciximab or similar antiplatelet agents in the previous 72 hours (Note that patients later found to have taken these medications will not be automatically excluded from the study.)
17. Use of sulfonylurea drugs within the prior 30 days
18. Treatment with another investigational drug within the prior 30 days
19. Allergy to sulfonylurea drugs
20. Known diagnosis of G6PD enzyme deficiency
21. PaO2 < 60 mm Hg on admission (for patients in whom blood gases are drawn per standard of care)
22. Non-English speaking legally authorized representative and subjects (University of Maryland only)
23. Prisoners or others who may be unable to make a truly voluntary and uncoerced decision whether or not to participate in the study
24. Any other clinical condition which in the opinion of the investigator makes the patient unsuitable for inclusion into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12-17 (Actual); Primary Completion 2015-02-20 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Edema | Baseline, Day 3, Day 90, and Day 180
  To be assessed using Magnetic Resonance Imaging (MRI).
Change from Baseline in Hemorrhage | Baseline, Day 3, Day 90, and Day 180
  To be assessed using MRI.
Number of Participants with Adverse Events and Serious Adverse Events | Up to 180 Days
  An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A serious adverse event is any AE that is fatal, life-threatening, requires or prolongs hospital stay, results in persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event

SECONDARY OUTCOMES:
Change from Baseline in Brain Volume | Baseline, Day 3, Day 90, and Day 180
  To be assessed using MRI.
Number of Participants with Abnormalities Associated with Brain Swelling | Baseline, Day 3, Day 90, and Day 180
  To be assessed using MRI and computed tomography (CT).
Change from Baseline in Glasgow Coma Scale (GCS) | Baseline up to Day 7
  The GCS is scored between 3 and 15 (3 = the worst, and 15 = best). It is composed of three parameters : Best Eye Response (scored on a scale of 1-4), Best Verbal Response (scored on a scale of 1-5), Best Motor Response (scored on a scale of 1-6)
Change from Baseline in Intracranial Pressure (ICP) | Baseline up to Day 7
Change from Day 30 in Extended Glasgow Outcome Scale (GOS-E) | Day 30, Day 60, Day 90, and Day 180
  The GOS-E assesses status in patients with traumatic brain injury on an 8-point scale. The minimum score is 1 and the maximum score is 8. The rating scale is as follows: 1- Dead, 2- Vegetative State, 3- Low Severe Disability, 4- Upper Severe Disability, 5- Low Moderate Disability, 6- Upper Moderate Disability, 7- Low Good Recovery, and 8- Upper Good Recovery
Number of Participants Requiring Decompression Craniectomy | Baseline up to Day 7
Number of Participants Experiencing Neuroworsening | Baseline up to Day 7
PK Parameter: Steady State Concentration of Glyburide | Baseline and 36 hours
Number of All-Cause and Neurological Mortalities | Up to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Remedy Pharmaceuticals
Locations (4):
- United States (4):
  - University of California, San Diego, San Diego, California
  - University of Maryland Medical Center, Shock Trauma Center, Baltimore, Maryland
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - VCU Medical Center, Richmond, Virginia